CLINICAL TRIAL: NCT06823557
Title: Gut2Brain: Investigation of the Mechanisms of the Gut-brain Axis in Binge Eating and Obesity
Brief Title: Investigation of the Mechanisms of the Gut-brain Axis in Binge Eating and Obesity.
Acronym: Gut2Brain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: University of Minho (Other); Braga Hospital (Unknown)
Responsible Party: Principal Investigator, Eva Conceição, Research Fellow, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPorto_Gut2Brain
Record Dates: First submitted 2025-01-17; First posted 2025-02-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: psychobiotic treatment; Study of neuro-psycho-biological mechanisms; Microbiota-Gut-Brain Axis (MGBA); Obesity; Binge eating disorder
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Prebiotics; Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) will compare three groups: a BED+obesity group, an obesity group (without BED), and a normal-weight group (without BED). Participants will be randomized and allocated into two arms in a double-blind, placebo-controlled design: an intervention group receiving a psychobiotic and a control group receiving a placebo matched in taste and appearance. Randomization will follow the CONSORT guidelines, utilizing a computer-generated sequence of random numbers in a 1:1 ratio. Groups will be matched based on BMI, age, and sex.
  Participants meeting the inclusion and exclusion criteria will undergo a semi-structured clinical interview to diagnose BED. They will also receive detailed information about the study and sign an informed consent form prior to participation. Assessments will take place at two time points: baseline (T0), before initiating the psychobiotic or placebo, and follow-up (T1), after completion of the assessment protocol.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychobiotic group (Experimental): An intervention group receiving a psychobiotic-a native inulin prebiotic. Native inulin extracted from chicory roots was selected as the psychobiotic since it is a mixture of short inulin molecules, which are metabolized primarily in the proximal colon and are more rapidly fermented, with longer chain ones, which are fermented later and slower in the distal colon. The psychobiotic nature of Inulin has been suggested in recent literature.
  Interventions: Dietary Supplement: Psychobiotic treatment
- Control group (Placebo Comparator): A control group receiving a taste/appearance-matched placebo- the maltodextrin. Maltodextrin is a carbohydrate consisting of short chains of glucose molecules. It is commonly used as a placebo in clinical trials, providing no significant health benefits or harm when consumed with moderation.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Psychobiotic treatment — The dietary supplementation will follow established guidelines, recommending an intake of 16 g of prebiotic per day, distributed across three meals, for a duration of 12 weeks.
  Other Names: Prebiotic; Inulin
  Arms: Psychobiotic group
Other: Placebo treatment — The control group will receive identical packaging that matches the experimental treatment in taste and appearance and will follow the same guidelines for consuming the placebo. For ethical reasons, after the end of the RCT, the control group will be given the option to receive the same prebiotic supplement.
  Other Names: Maltodextrin (Placebo)
  Arms: Control group

SUMMARY:
Binge Eating Disorder (BED) is a recently recognized eating disorder, characterized by recurrent episodes of overeating with a loss of control. Highly comorbid with obesity, BED is associated with poor outcomes in weight loss treatments and presents unique challenges due to its distinct neuro-psycho-biological mechanisms, which remain poorly understood. The Microbiota-Gut-Brain Axis (MGBA) is a bidirectional communication system linking the gut microbiota with the central nervous system, that plays a critical role in regulating appetite, mood, and eating behavior. Dysregulations in MGBA may contribute to the development and maintenance of BED, offering a novel framework for understanding its complex mechanisms and identifying new therapeutic targets. Psychobiotics -pre-, pro-, or symbiotics that modulate the microbiota- emerge as a promising treatment strategy to address BED symptoms by influencing MGBA activity.

The goal of this randomized clinical trial (RCT) is to investigate the role of psychobiotics in modulating the gut-brain axis and improving binge eating in adults, with a particular focus on evaluating these effects independently of obesity status. This project stands out for its comprehensive approach to understanding BED, integrating psychological, neurofunctional, hormonal, and microbiota factors that contribute to this complex disorder.

The main questions it aims to answer are:

* What specific alterations in the MGBA pathways are associated with BED?
* Can psychobiotic supplementation effectively reverse microbiota alterations and modulate MGBA activity, ultimately improving BED symptoms? Researchers will compare participants receiving psychobiotics to those receiving a look-alike substance that contains no drug (a placebo) to evaluate whether psychobiotics impact endocrine hormones, neurofunction, psychological and behavioral factors related to eating regulation, and BED symptoms.

Participants will:

* Undergo an assessment protocol that includes microbiota sampling, blood tests for hormone analysis, neurofunctional evaluations, and psychological/behavioral assessments before and after the psychobiotics/ placebo intervention.
* Take psychobiotics or a placebo daily for 12 weeks and receive well-being monitoring
* Participate in follow-up visits three months after the intervention to monitor changes in BED symptoms and related parameters.

DETAILED DESCRIPTION:
This research project aims to investigate the role of psychobiotics in reversing MGBA alterations specific to BED. Therefore, a two-arm Randomized Clinical Trial (RCT) will be conducted. Participants will include individuals with BED and obesity, individuals with obesity only, and individuals with normal weight that will be randomly assigned to one of two groups:

i) an intervention group receiving psychobiotic supplementation ii) a control group receiving placebo supplementation. The sample size was computed considering the sample needed for 3 groups comparison in the RCT. G Power was used for (Mixed) ANOVAs considering f = 0.25, power = 90%, α = 0.05, and corr = 0.5., and 15% dropout.

At both the beginning and end of the trial, participants will undergo an assessment protocol.

Assessment protocol:

Participants will be invited to visit Braga Hospital where the assessment will take place for a scheduled appointment to undergo the assessment protocol for approximately 2 hours. The first step will involve the assessment of appetitive hormones through blood samples collected at three time points. The first blood sample (0 minutes) will be taken after a 12-hour overnight fast. Participants will consume 600 mL of a standardized liquid test meal, and additional blood draws will occur 10 and 30 minutes after the meal.

Between the second and third blood samples collected, participants will respond with some self-report measures. Specifically, self-report measures will assess socio-demographic data (age, sex, gender, education levels, marital status, and weight history) and psychological aspects: 1) emotional regulation and impulse control, distress tolerance, and positive and negative affects; 2) eating behavior, assessing eating expectancy, emotional eating, compulsive eating, and restraint eating. Then participants will do resting-state functional magnetic resonance imaging (rs-FMRI) performed to evaluate resting-state network connectivity.

Stool samples will be collected using a kit that includes all the necessary tools for proper sample collection and preparation for microbiota analysis.

The psychobiotic and the placebo package and instructions will be delivered during this scheduled appointment in Braga Hospital. All participants will be contacted weekly during the 12-week trial to ensure/increase adherence to the guidelines of prebiotic/placebo intervention.

Statistical Analyses:

Overall, multivariate analysis of variance (MANOVA) and/or general linear models (GLM) with mixed-model repeated measures will be used to examine group differences related to MGBA mechanisms, as well as significant main effects and interaction effects between baseline (T0) and the end of the RCT (T1). Structural equation modeling (SEM) will be employed to evaluate MGBA mechanisms as mediators of the changes observed between T0 and T1.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese adults (25 with normal weight; 25 with obesity only (30 ≤ BMI < 40) and BED; 54 with BED)
* Residents in Portugal for the past 10 years

Exclusion Criteria:

* Significant weight loss (>5% of body weight) in the past 2 years
* Antibiotic use in the past 6 months
* History of surgery or medical/psychiatric diseases
* Pregnant or breastfeeding
* History of drug use or dependence
* Use of medications that impact weight
* Have metal implants or pacemakers

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota outcomes - Gut-Bacteria Composition | Change measures: baseline and end of treatment at 12 weeks
  Stool samples from each participant will be fermented by the prebiotic to allow direct comparison of individual alterations in vitro and in vivo of the microbiome. Changes in gut-bacteria composition and its adhesion into the mucus layer will be analyzed.
Gut Microbiota outcomes - Molecules released by the gut-bacteria | Change measures: baseline and end of treatment at 12 weeks
  Stool samples from each participant will be fermented by the prebiotic to allow direct comparison of individual alterations in vitro and in vivo of the microbiome. Molecules released by the bacteria, including short-chain fatty acids (SCFA), lipopolysaccharides (LPS), gamma-aminobutyric acid (GABA), dopamine, and serotonin, which modify host metabolism and central regulation of appetite directly via vagal stimulation or indirectly through immune-neuroendocrine mechanisms, will be traced during fermentations.
Psycho-behavioral outcomes - Three Factor Eating Questionnaire-21 | Change measures: baseline, end of treatment at 12 weeks and follow-up at 12 weeks post-treatment.
  Three Factor Eating Questionnaire-21 (TFEQ-21): assesses psychopathology and behaviors related to eating disorders, generating 3 subscales: emotional eating; compulsive eating; restraint eating.
Psycho-behavioral outcomes - Eating Expectancy Inventory | Change measures: baseline, end of treatment at 12 weeks and follow-up at 12 weeks post-treatment.
  - The Eating Expectancy Inventory (EEI): evaluates cognitive expectations regarding eating
Psycho-behavioral outcomes - Negative urgency subscale | Change measures: baseline, end of treatment at 12 weeks and follow-up at 12 weeks post-treatment.
  Negative urgency subscale from the Urgency, Premeditation, Perseverance, and Sensation Seeking scales (UPPS): assesses the tendency to act rashly/impulsively when experiencing negative emotions.
Psycho-behavioral outcomes - Difficulties in Emotion Regulation Scale | Change measures: baseline, end of treatment at 12 weeks and follow-up at 12 weeks post-treatment.
  Difficulties in Emotion Regulation Scale (DERS): self-report measure developed to assess difficulties in emotional dysregulation.
Psycho-behavioral outcomes - Distress Tolerance Scale | Change measures: baseline, end of treatment at 12 weeks and follow-up at 12 weeks post-treatment.
  The Distress Tolerance Scale (DTS): scale that assesses ability to experience, tolerate, and function in a context of emotional distress
Neurofunctioning outcomes - Default mode network | Change measures: baseline and end of treatment at 12 weeks
  Neurofunctioning will be assessed through rs-fMRI. Specifically, we aim to compare the resting-state networks (RSNs), such as the default mode network (DMN), the salience network (SN), the meso/paralimbic network (MPN), and the executive network (EN) across the three groups. The DMN is involved in self-referential processing, which includes monitoring the external environment as well as physical and emotional states.
Neurofunctioning outcomes - Salience network | Change measures: baseline and end of treatment at 12 weeks
  Neurofunctioning will be assessed through rs-fMRI. Specifically, we aim to compare the resting-state networks (RSNs), such as the default mode network (DMN), the salience network (SN), the meso/paralimbic network (MPN), and the executive network (EN) across the three groups. The DMN is involved in self-referential processing, which includes monitoring the external environment as well as physical and emotional states. The SN is involved in detecting the salience of stimuli, integrating emotional arousal, food, and reward processing.
Neurofunctioning outcomes - Meso/Paralimbic network | Change measures: baseline and end of treatment at 12 weeks
  Neurofunctioning will be assessed through rs-fMRI. Specifically, we aim to compare the resting-state networks (RSNs), such as the default mode network (DMN), the salience network (SN), the meso/paralimbic network (MPN), and the executive network (EN) across the three groups. The MPN is involved in processing emotional information and interoceptive awareness.
Neurofunctioning outcomes - Executive network | Change measures: baseline and end of treatment at 12 weeks
  Neurofunctioning will be assessed through rs-fMRI. Specifically, we aim to compare the resting-state networks (RSNs), such as the default mode network (DMN), the salience network (SN), the meso/paralimbic network (MPN), and the executive network (EN) across the three groups. The EN is involved in cognitive control and inhibitory processes, such as the termination of food consumption
Appetitive hormones outcomes - Ghrelin | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  * Ghrelin is an orexigenic hormone with stimulatory effects on appetite and food intake.
Appetitive hormones outcomes - Glucagon-Like Peptide 1 | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  * Glucagon-Like Peptide 1 (GLP-1) have an anorexigenic effect and are thought to contribute to impaired satiation and binge eating tendencies. GLP-1 has been the target of novel therapeutics for weight loss, but few studies have examined its impact on BED.
Appetitive hormones outcomes - Peptide YY | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  - Peptide YY (PYY) have an anorexigenic effect and are thought to contribute to impaired satiation and binge eating tendencies.
Appetitive hormones outcomes - Leptin | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  * Leptin acts as a regulatory signal reflecting the adipose tissue stores. Both insufficiency and resistance to its actions promote hunger and increased food intake. Leptin can decrease food reward and act in the central nervous system as regulators of energy homeostasis.
Appetitive hormones outcomes - Insulin | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  Insulin can decrease food reward and act in the central nervous system as regulators of energy homeostasis.
Appetitive hormones outcomes - Cortisol | Change measures: baseline and end of treatment at 12 weeks
  Assessment of appetitive hormones that modulate eating behavior:
  - Cortisol is responsible for the stress response, acting on the hypothalamic-pituitary axis, and it is associated with increased eating

SECONDARY OUTCOMES:
Eating Disorder Examination | baseline moment
  Eating Disorder Examination (EDE): semi-structured clinical interview for the diagnosis of binge eating disorder

CONTACTS AND LOCATIONS:
Overall Officials: Eva M. Conceição, Principal Investigator — Center for Psychology at University of Porto (CPUP); Clarisse N. Salomé, Principal Investigator — Center for Engineering Biological (CEB) at University of Minho
Locations (1):
- Center for Psychology at University of Porto, Porto, Paranhos, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from jan 2030 to jan 2035
Access Criteria: Researcher with research track record in the filed by contacting the PI of the study.